CLINICAL TRIAL: NCT03384017
Title: The Impact of Transcutaneous Spinal Cord Stimulation (TSCS) and Gait Training on Walking Function in Patients With Spinal Cord Injury
Acronym: TSCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Rebecca Martin, OTR/L, OTD, Manager Clinical Education and Training, International Center for Spinal Cord Injury Assistant Professor, Johns Hopkins School of Medicine, Dept. of Physical Medicine and Rehabilitation, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00053916
Record Dates: First submitted 2017-12-12; First posted 2017-12-27 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All assessors will be blind to intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TSCS and gait training (Experimental)
  Interventions: Other: Transcutaneous Spinal Cord Stimulation and Gait Training

INTERVENTIONS:
Other: Transcutaneous Spinal Cord Stimulation and Gait Training — TSCS will be applied using a midline electrode placed on the skin between spinous process T11 -T12 and two electrodes placed symmetrically on the skin over the lower abdomen as anodes. A symmetrical biphasic rectangular waveform, at 50 Hz and 1 millisecond, is used to provide 30 continuous minutes of stimulation.
  Subjects will participate in 24 two-hour sessions of physical therapy over eight weeks. In each session, subjects will receive TSCS continuously for 30 minutes, using the parameters outlined above. During stimulation, subjects will participate in strengthening, segmental task practice, and gait-based interventions. Participation in gait training will continue following the stimulation period for the duration of the session.

SUMMARY:
Aim 1: Determine the neurophysiologic impact of Transcutaneous Spinal Cord Stimulation (TSCS) within a single session. The investigators hypothesize that subjects will demonstrate increased volitional muscle activity and strength with TSCS. This will be assessed by surface EMG and hand-held dynamometry of the dominant-side quadriceps muscle during maximum volitional contraction (MVC) and measurement of gait speed. Subjects will be tested in both TSCS and sham conditions.

Aim 2: Determine the impact of TSCS and gait training on walking function. The investigators hypothesize that concurrent TSCS and gait training will augment walking function in subjects with iSCI, as compared to gait training alone. Subjects will participate in an eight-week program of gait training with TSCS and be assessed with clinically relevant outcome measures, to include the Timed Up and Go, 10-Meter Walk Test, Walking Index for Spinal Cord Injury II, and 6-Minute Walk Test.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* >1 year post SCI
* Non-progressive SCI
* Neurological level above T10
* Tolerates upright position for >30 minutes
* Medically stable (no hospitalizations in last 3 months)
* Able to comply with procedures and follow up
* Are legally able to make their own health care decisions

Exclusion Criteria:

* Progressive SCI/D (MS, ALS, ADEM, etc.)
* Open wounds at stimulation site
* Pregnant women
* ROM limitations impacting gait training
* Cardiac pacemaker/defibrillator
* Active cancer diagnosis
* Currently receiving TSCS
* Evidence of uncontrolled autonomic dysreflexia
* Non-English speaking subjects will not be targeted

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Change in walking speed | at the start, week 4, and week 8
  10-Meter Walk Test

SECONDARY OUTCOMES:
Change in walking capacity | at the start, week 4, and week 8
  Timed Up and Go
Change in level of assistance and assistive device for walking | at the start, week 4, and week 8
  Walking Index for Spinal Cord Injury II
Change in walking endurance | at the start, week 4, and week 8
  6-Minute Walk Test

CONTACTS AND LOCATIONS:
Locations (1):
- Rebecca Martin, OTR/L, OTD, CPAM, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No